CLINICAL TRIAL: NCT05950204
Title: Effect of Combined Supplementation With Long-chain ω-3 Polyunsaturated Fatty Acids, Vitamin D, and Calcium as a Potential Adjuvant in the Preservation of Bone Mass and Bone Turnover Biomarkers in Patients With Acute Lymphoblastic Leukemia.
Brief Title: Effect of Supplementation With ω-3 Fatty Acids, Vitamin D and Calcium in Patients With Acute Lymphoblastic Leukemia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, María de Lourdes Barbosa Cortés, Associated researcher, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2019-785-021
Record Dates: First submitted 2023-07-05; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Acute Lymphoblastic Leukemia; Vitamin d Deficiency
Keywords: Acute Lymphoblastic Leukemia; Bone Turnover Biomarkers; Corticosteroids; Bone Mineral Density; Long-Chain polyunsaturated fatty acids; n-3 fatty acids; Vitamin D
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Vitamin D Deficiency | interventions — Vitamin D; Cholecalciferol; Calcium; Calcium Carbonate

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): 100 mg/kg/d of LCPUFA-ω3 with a ceiling dose of 3 g/d, + 1,000 mg of calcium/day and 4,000 IU (100 µg)/d of VD in those children > 9 years and 20,000 UI/week = 2,857 UI/d in those < 8 years for 6 weeks
  Interventions: Dietary Supplement: ω-3 polyunsaturated fatty acids (DHA and EPA), Vitamin D (cholecalciferol), Calcium (calcium carbonate)
- Group B (Active Comparator): 1,000 mg of calcium/day and 4,000 IU (100 µg)/d of VD in those children > 9 years and 20,000 UI/week = 2,857 UI/d in those < 8 years for 6 weeks
  Interventions: Dietary Supplement: ω-3 polyunsaturated fatty acids (DHA and EPA), Vitamin D (cholecalciferol), Calcium (calcium carbonate)

INTERVENTIONS:
Dietary Supplement: ω-3 polyunsaturated fatty acids (DHA and EPA), Vitamin D (cholecalciferol), Calcium (calcium carbonate) — Intervention with 100 mg/kg/d of LCPUFA-ω3 with a ceiling dose of 3 g/d, + 1,000 mg of calcium/day and 4,000 IU (100 µg)/d of VD in those children > 9 years and 20,000 UI/week = 2,857 UI/d in those < 8 years for 6 weeks. The other group of patients will receive only the same dose of VD and calcium.
  Other Names: LCPUFA-ω3; Vitamin D; Calcium

SUMMARY:
The purpose of this study is to evaluate the efficacy of supplementation with Omega 3, Vitamin D and Calcium, in a cohort of children with ALL undergoing treatment and compare changes in the concentrations of biomarkers of bone resorption (TRAP5b, CTX, and RANKL), the RANKL/OPG ratio, and biomarkers of bone formation (BALP, OC, PINP, PICP and OPG) after 6 and 12 weeks of supplementation.

DETAILED DESCRIPTION:
In pediatric hematological patients, the administration of high and prolonged doses of corticosteroids has a negative effect on bone metabolism, causing a significant reduction in bone mineral density (BMD). Maintaining adequate levels of vitamin D (VD) and calcium is crucial for bone health, and deficiencies in these nutrients increase the risk of osteoporosis. Children with acute lymphoblastic leukemia (ALL) have been found to have a high prevalence of VD deficiency. Bone turnover markers (BTMs) are substances produced by osteoblasts and osteoclasts that provide information about the dynamic remodeling of bone. Limited research has investigated the role of BTMs in pediatric ALL patients receiving VD supplementation.

Emerging evidence suggests that long-chain ω-3 polyunsaturated fatty acids (LCPUFA-ω3) play a significant role in bone health. Consumption of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) may inhibit bone resorption and promote bone formation in humans.

Currently, there are no randomized controlled clinical trials comparing the effects of combined supplementation with LCPUFA-ω3, VD, and calcium on BTMs in children with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Children with acute lymphoblastic leukemia in maintenance
* authorization from both parents or legal guardian for recruiting of the child into the study with consent have been explained
* Must be able to swallow capsules

Exclusion Criteria:

* Patients with acute or chronic renal failure
* Added pathology
* Fish Hypersensitivity
* Down´s Syndrome

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-09-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Vitamin D status and changes in the concentrations of biomarkers of bone resorption | at the time of the recruitment, 6 weeks of supplementation and after 6 weeks without supplementation
  After 6 weeks of supplementation, VD (1-25 hydroxyvitamin D) levels will be evaluated by liquid chromatography coupled to high-resolution mass spectrometry (Waters Acquity UPLC H-Class). The biomarkers of BTMs will be analyzed by ELISA. Parathormone, phosphorus and calcium will be assessed by spectrophotometry, and 3 LCPUFA-ω3 will be analyzed by gas chromatography.

SECONDARY OUTCOMES:
Concentrations of inflammatory markers (IL-6 and TFN) | at the time of the recruitment, 6 weeks of supplementation and after 6 weeks without supplementation
  changes in the concentrations of inflammatory markers (IL-6 and TFN) in a cohort of children with ALL undergoing treatment after 3 months of supplementation with LCPUFA-ω3, VD, and calcium compared to a group receiving only calcium and VD

CONTACTS AND LOCATIONS:
Overall Officials: María de Lourdes Barbosa Cortés, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Unit of research in Nutrition, Pediatric Hospital, Instituto Mexicano del Seguro Social, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No